CLINICAL TRIAL: NCT02675322
Title: Effects of Danlou Tablets to Prevent Left Ventricular Remodeling After Myocardial Infarction: A Double-blind, Randomized, Placebo Controlled, Pilot Study
Brief Title: Danlou Tablets to Prevent Left Ventricular Remodeling
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: shuai Mao (Other)
Responsible Party: Sponsor-Investigator, shuai Mao, Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangdong Provincial Hospital of Traditional Chinese Medicine
Organization: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GuangdongPHTCM
Record Dates: First submitted 2016-02-01; First posted 2016-02-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Left Ventricular Remodeling; Acute Myocardial Infarction
MeSH Terms: conditions — Ventricular Remodeling | interventions — danlou tablet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Danlou Tablets (Experimental): Danlou tablets (4.5 g oral dose taken once daily) for 90 days
  Interventions: Drug: Danlou Tablets
- placebo (Placebo Comparator): matching placebo for 90 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Danlou Tablets — Danlou tablets were approved by China Food and Drug Administration for the treatment of ischemic heart disease in 2005 (Z20050244).
  Other Names: Danlou
  Arms: Danlou Tablets
Other: Placebo — Placebo with no chemical effects.
  Arms: placebo

SUMMARY:
Danlou tablets are Chinese patent medicine which has been approved in China for the treatment of ischemic heart disease, but the evidence supporting its efficacy on cardiac remodeling remains unclear. This pilot study was designed to determine whether Danlou tablets reduced adverse left ventricular (LV) remodeling in patients with acute myocardial infarction (MI). Patients following acute MI were enrolled and randomly allocated to Danlou tablets (4.5 g q.d. for 90 days) or placebo, superimposed on standard medications for the treatment of MI. Major end points were changes in LV volumes and ejection fractions as evaluated by serial echocardiography in addition to clinical outcomes were also determined.

DETAILED DESCRIPTION:
This randomized, prospective, double-blind, placebo-controlled, parallel-group clinical trial was performed in two institutions (Guangdong Provincial Hospital of CM and Wuyi Hospital of CM). The study was conducted in accordance with the Declaration of Helsinki and its text revisions and all participants provided written informed consent before enrollment. The Clinical Research Ethical Committee at Guangdong Provincial Hospital of Chinese Medicine approved the research protocol (B2011-41-01).

Once eligible candidates had undergone PCI, they were admitted to the coronary intensive care unit and received standard treatment according to the institutional protocol based on American College of Cardiology/ American Heart Association and European Society of Cardiology guidelines.20 Simultaneously, patients were randomized assigned in a 1:1 ratio to receive Danlou tablets (4.5 g oral dose taken once daily) or matching placebo for 90 days according to a computer-generated site-stratified, block randomization schedule. Danlou tablets were approved by China Food and Drug Administration for the treatment of ischemic heart disease in 2005 (Z20050244).

ELIGIBILITY:
Inclusion Criteria:

* acute myocardial infarction
* successfully underwent revascularization

Exclusion Criteria:

* previous myocardial infarction within 30 days
* malignant arrhythmia
* congenital heart disease
* cardiac shock
* documented or suspected history of heart failure or depressed LV ejection fraction <15%
* planned coronary artery bypass grafting
* a life expectancy of <1 year
* hepatic impairment
* glomerular filtration rate ≤30 mL/min per 1.73 m2
* autoimmune or connective tissue disease
* chronic substance abuse or psychiatric illness
* unable to complete 3 month clinical follow-up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
change in the Left Ventricular End Diastolic Volume Index from baseline to 90 days | 90 days
  Left Ventricular End Diastolic Volume Index (LVEDVi) measured by two-dimensional echocardiography.

SECONDARY OUTCOMES:
changes in Left ventricular End Systolic Volume Index from baseline to 90 days | 90 days
  Left Ventricular End Systolic Volume Index (LVESVi) measured by two-dimensional echocardiography.
Major adverse cardiovascular events | 90 days
  Major adverse cardiovascular events includes cardiac death, cardiac shock, myocardial infarction, documented unstable angina requiring revascularization (bypass surgery or repeat PCI), severe angina or severe heart failure.
adverse events | 180 days
Left ventricular Ejection Fraction from baseline to 90 days | 90 days
  Left ventricular Ejection Fraction (LVEF) measured by two-dimensional echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: minzhou zhang, M.D., Study Chair — Heart Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mao S, Wang L, Ouyang W, Zhou Y, Qi J, Guo L, Zhang M, Hinek A. Traditional Chinese medicine, Danlou tablets alleviate adverse left ventricular remodeling after myocardial infarction: results of a double-blind, randomized, placebo-controlled, pilot study. BMC Complement Altern Med. 2016 Nov 8;16(1):447. doi: 10.1186/s12906-016-1406-4. PMID 27825334